CLINICAL TRIAL: NCT06995196
Title: The Effect of the Use of ReLiver-N App Developed for Patients With Liver Cirrhosis on Hepatic Rehabilitation: A Randomized Controlled Single-Blind Study
Brief Title: Care Algorithm and Clinic Decision System on Hepatic Rehabilitation in Patients With Liver Cirrhosis
Acronym: ReLiver-NApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ferya Celik, Research Assistant Dr, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TÜBİTAK 123S032; 123S032 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Liver Cirrhosis
Keywords: nursing care; hepatic rehabilitation; care algorithm; patient activation; patient clinic decision system; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Patient Participation | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group access all the content of ReLiver-N App incluiding educational content, patient activation intervensions, care algorithms, and patient clinical decision systems.
  Interventions: Behavioral: ReLiver-N App
- Active Control (Active Comparator): Patients in the active control group access only education content of ReLiver-N App and patient activation intervention without feedback of their results.
  Interventions: Behavioral: ReLiver-N App

INTERVENTIONS:
Behavioral: ReLiver-N App — Intervention for intervention group: Patients will access all content of ReLiver-N App. The ReLiver-N App has comprehensive health education, patient activation practices, care algorithm, and clinical decision system, to provide and maintain the hepatic rehabilitation of patients with liver cirrhosis and to evaluate the effect of the use of ReLiver-N App on hepatic rehabilitation. Care algorithm and clinical decision system will be evaluated results of patient activation as "normal", "controllable", "urgent". Feedbacks will be sent to patients based on the evaluations.
  Other Names: Intervention for active control gorups: Patients in the active control groups will access only health education content of ReLiver-N App

SUMMARY:
Liver cirrhosis is an important public health problem that causes morbidity and mortality. In order to provide hepatic rehabilitation of patients with liver cirrhosis, interventions that provide active care practices by patients and evaluation of results are needed. In this trial, it is aimed to develop a nurse-led mobile health application (ReLiver-N App- Rehabilitation of Liver by Nurse), which has comprehensive health education, patient activation practices, care algorithm, and clinical decision system, to provide and maintain the hepatic rehabilitation of patients with liver cirrhosis and to evaluate the effect of the use of ReLiver-N App on hepatic rehabilitation. Care algorithm and clinical decision system will be evaluated results of patient activation as "normal", "controllable", "urgent". Feedbacks will be sent to patients based on the evaluations. This project consists of two phases, methodological and randomized controlled experimental study. The first stage, in which ReLiver-N App will be developed, is planned as a methodological study, and the second stage, in which the effect of ReLiver-N App on hepatic rehabilitation will be evaluated, as a randomized controlled single-blind experimental study. ReLiver-N App will be developed in line with the steps of the Design Based Research Model. The sample size of the project is planned to consist of 56 patients with liver cirrhosis. Patients with a diagnosis of liver cirrhosis, 18 years of age and older, with the severity of the disease in Child Pugh A and B categories, without verbal or written communication barriers, with a smart phone, and who consented to participate in the study will constitute the sample. Pre-tests will be applied by face-to-face interview method. Assignment of patients to intervention and control groups will be made by block randomization. While patients in the intervention group access all the content of ReLiver-N App; patients in the control group will not have access to any data on the intervention. It is planned that the project will be implemented for 90 days and follow up evaluations will be made every month. Follow up assessments and post-test data will be available online via the ReLiver-N App. The dependent variable of the project is hepatic rehabilitation, and the independent variable is ReLiver-N Intervention Protocol.

DETAILED DESCRIPTION:
Liver cirrhosis, a progressive, chronic disease characterized by fibrotic tissue, regenerative nodules, and loss of function in liver cells, is an important public health problem that causes morbidity and mortality. The European Association for the Study of the Liver (EASL) recommends providing appropriate treatment and care at an early stage, preventing the development of complications, and early recovery in order to reduce morbidity and mortality due to liver cirrhosis. In line with this recommendation, treatment and care practices in patients with liver cirrhosis should be planned to prevent the development and recurrence of life-threatening symptoms and to help improve them. It is stated that hepatic rehabilitation programs to be developed for patients with liver cirrhosis are an important part of achieving this goal. Hepatic rehabilitation includes practices carried out to maintain and improve the health of hospitalized or discharged liver cirrhosis patients, to ensure the active participation of patients in self-care practices, to prevent and improve complications, and to provide palliative care when necessary. Hepatic rehabilitation programs that patients can access continuously, use as a source of information about their diseases, learn and apply care practices, and receive instant feedback in line with real-time health data are needed for hepatic rehabilitation. In this trial, the ReLiver-N Intervention Protocol was created to provide hepatic rehabilitation for patients diagnosed with liver cirrhosis. The content of the ReLiver-N Intervention Protocol consists of comprehensive health education, patient activity practices (daily patient activity practices: medication use, weight monitoring, edema monitoring, intake-exit monitoring, defecation monitoring; weekly patient activity practices: fever, blood pressure, pulse measurement), care algorithms, and patient decision support system. The ReLiver-N Intervention Protocol is being developed within the scope of the Design-Based Research Method.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with liver cirrhosis Had Child-Pugh A and B categories 18 years of age or older No barriers to verbal or written communication Having internet at home and a smartphone Patients who consented to participate in the study.

Exclusion Criteria:

Had Child-Pugh C category Had pregnant Liver transplanted Diagnosed with hepatocellular carcinoma Having dementia Having been diagnosed with a psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Patient Activation-Patient Activation Measure | 12 weeks
  The Patient Activation Measure (PAM) is a 13-item measure that assesses patient knowledge, skill, and confidence for self-management. The higher score showes better outcome.
Self-efficacy, Self-efficacy for Managing Chronic Disease 6-item Scale | 12 weeks
  This 6-item scale contains items taken from several SE scales developed for the Chronic Disease Self Management study. The higher score showes better outcome.
Quality of life - Chronic Liver Disease Questionnaire | 12 weeks
  The CLDQ includes 29 items in the following domains: abdominal symptoms, fatigue, systemic symptoms, activity, emotional function and worry. The higher score showes better outcome.

SECONDARY OUTCOMES:
Hospital readmissin | 12 weeks
  Hospital readmissions frequently occur in patients with cirrhosis and are associated with liver disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ferya Celik, PhD, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It could be shared on demand
Supporting Information: Study Protocol
Time Frame: 2 years after the article was published
Access Criteria: It could be shared on demand